CLINICAL TRIAL: NCT06514885
Title: Influence of Silver Diamine Fluoride Application on the Restorative Treatment for Root Caries
Brief Title: Silver Diamine Fluoride Application on Root Caries Fillings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW23-005
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Root Caries
Keywords: silver diamine fluoride; older adults; restorative treatment; root caries
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Intervention Model Description: two-arm randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, operators and investigators will not be informed of the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDF group (Experimental): Participants of SDF group will be applied with SDF before placement of root caries restoration
  Interventions: Other: SDF solution application
- Control group (Placebo Comparator): Participants of control group will be applied with placebo (tonic water) before placement of root caries restoration
  Interventions: Other: Tonic water

INTERVENTIONS:
Other: SDF solution application — silver diamine fluoride (SDF) solution is highly effective in stopping and arresting the progress of decay in dental roots of older adults. The American Dental Association (ADA) has published a guideline based on the up-to-date evidence to support the use of SDF for managing tooth decay. As a non-invasive procedure, application of SDF is simple, quick, painless and non-aerosol generated.
  Arms: SDF group
Other: Tonic water — Tonic water will be used as a placebo to mimic the SDF solution.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn the influence of prior silver diamine fluoride (SDF) application on root caries fillings.

The main questions to answer

1. Compare the success of fillings placed in dental root decay that have prior SDF application and those without prior SDF application;
2. Compare patient-based subjective evaluations on the two approaches mentioned above in treating root caries.

Participants will be allocated into two group

1. prior SDF application before receiving root caries fillings
2. directly receiving root caries fillings without any SDF application

DETAILED DESCRIPTION:
The aim of the proposed study is to investigate the influence of prior SDF application on the restorative treatment of root caries.

The objectives of the study are to

1. Compare the success rate of restorations placed in root caries lesions that have prior SDF application and that of restorations placed without prior SDF application;
2. Compare patient-based subjective evaluations on the two different approaches mentioned-above in treating root caries lesions.

Hypotheses to be tested:

1. Prior SDF application increases the success rate of restorations placed in root caries;
2. Patient-based subjective evaluations of the treatment outcomes are better when SDF is applied to the root caries lesions prior to restoring the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (aged 60 or above)
* At least one untreated decayed dental root

Exclusion Criteria:

* No self-care ability for basic daily activities
* Teeth with severe decay (cannot be filled)
* Teeth indicated for extraction

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 24 months follow-up
  Compare the success rate of restorations placed in root caries lesions that have prior SDF application or that of restorations placed without prior SDF application

SECONDARY OUTCOMES:
Patient-based subjective evaluation | 24 months follow-up
  Compare patient-based subjective evaluations on the two different approaches in treating root caries lesions.
  The Chinese version of General Oral Health Assessment Index (GOHAI) will be adopted as a tool to assess the oral health-related quality of life (OHRQoL) of the participants. It contains 12 questions covering three domains: physical function, pain and discomfort, and psychosocial function. The total GOHAI score is generated by adding up the score of each response to the 12 questions, and the total score ranges from 12 to 60. A higher score indicates a better perceived OHRQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li R, Lo EC, Liu BY, Wong MC, Chu CH. Randomized clinical trial on arresting dental root caries through silver diammine fluoride applications in community-dwelling elders. J Dent. 2016 Aug;51:15-20. doi: 10.1016/j.jdent.2016.05.005. Epub 2016 May 18. PMID 27208876
- [Background] Zhang W, McGrath C, Lo EC, Li JY. Silver diamine fluoride and education to prevent and arrest root caries among community-dwelling elders. Caries Res. 2013;47(4):284-90. doi: 10.1159/000346620. Epub 2013 Feb 5. PMID 23392087
- [Background] Lo EC, Luo Y, Tan HP, Dyson JE, Corbet EF. ART and conventional root restorations in elders after 12 months. J Dent Res. 2006 Oct;85(10):929-32. doi: 10.1177/154405910608501011. PMID 16998134

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT06514885/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT06514885/ICF_001.pdf